CLINICAL TRIAL: NCT02955264
Title: Using D-Galactose as a Food Supplement in Congenital Disorders of Glycosylation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-517339
Record Dates: First submitted 2016-09-14; First posted 2016-11-04 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Congenital Disorders of Glycosylation
Keywords: Glycosylation; Glucose Metabolic Disorder; Galactose
MeSH Terms: conditions — Congenital Disorders of Glycosylation; Glucose Metabolism Disorders | interventions — Galactose

STUDY DESIGN:
Intervention Model Description: Dietary Supplement: D-Galactose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-Galactose (Experimental): D-Galactose is an oral powdered supplement to be taken by mouth. For the first 6 weeks galactose will be given at the dose 0.5g per kg, then from weeks 7-12 at 1.0g per kg, lastly from weeks 13 to 18 at 1.5g per kg (with a maximum daily dose of 50g).
  Interventions: Dietary Supplement: D-Galactose

INTERVENTIONS:
Dietary Supplement: D-Galactose — D-Galactose is an oral powdered dietary supplement to be taken by mouth.

SUMMARY:
The goal of this study is to better characterize the metabolic alterations and sugar structure alterations (glycosylation abnormalities) in patients diagnosed with Congenital Disorders of Glycosylation. The investigators aim to assess the safety and tolerability of oral galactose treatment in a small pilot group of Congenital Disorders of Glycosylation patients. The investigators will also determine the relationship between simple milk sugar intake (galactose dose) in the diet and the blood and urine markers of protein glycosylation abnormalities.

DETAILED DESCRIPTION:
The primary hypothesis in this study is that adding simple milk sugar (galactose) to the diet of Congenital Disorders of Glycosylation patients will normalize the metabolic abnormalities. The secondary hypothesis posits that galactose intervention in Congenital Disorders of Glycosylation patients will normalize specific physiological biomarkers of protein glycosylation that can be utilized for future phase II/III trial development. The knowledge gained from the investigation of these two aims will help the investigators learn more about the disrupted metabolic mechanism of this disease and should lead to the identification of new disease biomarkers that can be used to evaluate clinical efficacy in future therapeutic trials.

Over a two-year period, the investigators will enroll patients diagnosed with Congenital Disorders of Glycosylation. The investigators propose to administer oral galactose supplementation for a period of 18 weeks in increasing dose to assess its effectiveness at normalizing glycosylation. Galactose will be given in a series of doses within the range of normal dietary intake of galactose over fixed time points. To assess the effects of oral galactose supplementation for each participant, changes in participant growth, as well as blood sugar levels, coagulation parameters and liver function (the primary clinical features of Congenital Disorders of Glycosylation) will be correlated with biomarkers derived from participant blood and urine samples obtained at key time points and then compared to standard normative ranges of data for each measure.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically and genetically proven Congenital Disorders of Glycosylation.

Exclusion Criteria:

* Any of the following conditions:
* Aldolase B Deficiency
* Galactosemia (unable to process galactose)
* Hemolytic uremic syndrome
* Severe anemia
* Diagnosis of intellectual disability or developmental delay
* Galactose Intolerance
* Has previously experienced any of the following severe side effects from oral galactose:
* Diarrhea
* Vomiting
* Constipation
* Galactosuria (Galactose in the urine)
* Increased liver glycogen storage.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Metabolic Function | 18 weeks
  Assess if the introduction of galactose into the subject's diet will normalization metabolic function. Metabolic function will be based on liver function and used for muscle enzyme tests, thyroid and growth hormone measurement, coagulation and anti-coagulation factors, blood sugar and milk-acid and biochemical/metabolic parameters. These measurements will be assessed together to see how many subjects will remain with abnormal values or change to within normal levels.

SECONDARY OUTCOMES:
Biomarkers for protein glycosylation | 18 weeks
  Identify potential biomarkers for glycosylation and metabolic dysfunction. And learn the physiological effect of adding galactose to the diet on known biomarkers for protein glycosylation. Specific biomarkers that will be examined include: transferrin glyco isoforms, antithrombin III, coagulation factor IX and XI, IGFBP3 and TSH. These measurements will be assessed together to see how many subjects will remain with abnormal values or change to within normal levels.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Morava-Kozicz, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Witters P, Andersson H, Jaeken J, Tseng L, van Karnebeek CDM, Lefeber DJ, Cassiman D, Morava E. D-galactose supplementation in individuals with PMM2-CDG: results of a multicenter, open label, prospective pilot clinical trial. Orphanet J Rare Dis. 2021 Mar 20;16(1):138. doi: 10.1186/s13023-020-01609-z. PMID 33743737